CLINICAL TRIAL: NCT04142996
Title: A Naturalistic Study Comparing Uni- and Bi-lateral Theta Burst Stimulation in Major Depression
Brief Title: Comparing Uni- and Bi-lateral TBS in Major Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Ottawa Mental Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019017
Record Dates: First submitted 2019-10-15; First posted 2019-10-29 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Major Depressive Episode

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both participants and research team members conducting the interviews and the TBS treatment will be blinded to the TBS treatment condition. In the unilateral arm, the right-sided stimulation will be applied with the placebo side of the coil. In the bilateral arm, the right-sided stimulation will be applied with the active side of the coil. As such, all participants will receive a total of 4 minutes of daily TBS. The master randomization list was created by a scientist of the research centre that is not involved in the research project.
  The patient's study identification (ID) code is entered into the device and a software-controlled switch then automatically selects the active or the sham coil for stimulation. The electronic positioning sensor built in the coil for monitoring the coil orientation checks against the entered patient's study ID and will enable the device and start the treatment procedure only if the coil orientation is matching the patient's study ID value.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unilateral TBS (Active Comparator): Intermittent Theta Burst Stimulation (iTBS) will be applied to the left DLPFC. Realistic sham continuous TBS (cTBS-sham) will be applied to the right DLPFC. Participants will receive daily sessions (Mon-Fri) for 4 to 6 weeks (stop at 4 weeks if remission is achieved).
  Interventions: Device: Theta burst stimulation
- Bilateral TBS (Active Comparator): Intermittent Theta Burst Stimulation (iTBS) will be applied to the left DLPFC and continuous TBS (cTBS) will be applied to the right DLPFC. Participants will receive daily sessions (Mon-Fri) for 4 to 6 weeks (stop at 4 weeks if remission is achieved).
  Interventions: Device: Theta burst stimulation
- Maintenance Phase: Flexible (Active Comparator): The flexible maintenance protocol will be based on symptom emergence. Participants will receive a fixed TBS (2x/week) schedule for the first month. For the following months (2-6), they will come in for an assessment (HRSD-17) to determine how many TBS sessions (0, 1, or 2) they receive on a flexible basis.
  Interventions: Device: Theta burst stimulation

INTERVENTIONS:
Device: Theta burst stimulation — Cool B70 coil (left DLPFC) and Cool B65 active/placebo coil (right DLPFC), with X100 MagPro rTMS Device (Magventure A/S, Farum, Denmark)

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) is a Health Canada approved treatment for major depression. Theta burst stimulation (TBS) is a very promising new treatment for major depression that allows a 15-fold reduction in duration of daily sessions. However, no large scale naturalistic study has assessed the superiority of bilateral TBS in comparison with unilateral left TBS. In fact, no TBS study thus far has included both unipolar and bipolar depression, or other psychiatric comorbidities such as anxiety. Maintenance has yet to be studied with TBS, along with an effective maintenance protocol to prevent relapse. Our study aims to explore and address these gaps.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is a Health Canada approved treatment for major depression. Typical treatments involve 30 to 45 minutes daily session delivered over 4 to 6 weeks. Recent technical advances allowed the development of theta burst stimulation (TBS), a novel rTMS paradigm which reduces daily sessions to 3 to 4 minutes while maintaining the same clinical efficacy. However, it remains to be determined if applying TBS to both sides of the frontal cortex (i.e. bilateral TBS) is more efficient than delivering it to only one side (i.e. unilateral TBS). In addition, it is difficult to predict treatment response as there is a lack of tools to identify potential responders early on in the treatment phase. Finally, the effects of rTMS are known to last up to 12 months after the treatment. To avoid relapse, a maintenance phase is typically introduced after treatment in which treatment sessions are delivered at a gradually decreasing rate. This study proposes to bridge these gaps by conducting a randomized double-blinded naturalistic superiority trial in which the efficacy of bilateral and unilateral TBS will be compared in individuals with a diagnosis of major depressive episodes. Neurobiological markers of response will be assessed at different time points. In people that respond to treatment, a 6-month maintenance phase will be conducted using a flexible schedule.

The study has four primary aims:

1. To compare the efficacy of bilateral and unilateral TBS on symptoms of depression, as well as rates of remission and response
2. To investigate how unilateral and bilateral TBS modulates brain activity in the dorsolateral prefrontal cortex (DLPFC) using interleaved TMS-EEG
3. To investigate neural predictors of the clinical response to TBS.
4. To assess the efficacy of a flexible schedule of maintenance on a period of 6 months on symptoms of depression and rate of relapse.

TREATMENT PHASE TBS treatment will be administered 5 days/week (on weekdays) over a first phase of 4 weeks (20 sessions). If remission is achieved (Hamilton Rating Scale for Depression-17 score < 8), treatment will cease and the patient will move on to the maintenance phase. Non-remitters will receive a second phase of treatment, consisting of an additional 2 weeks (10 sessions, for a total of 30). After 6 weeks, all responders may move on to the maintenance phase.

MAINTENANCE PHASE The maintenance phase will be of 6 months duration from the end of the randomized treatment. For each TBS condition, responders will be assigned to a flexible maintenance protocol based on symptom emergence. Participants will receive a fixed 2x/week schedule for the month 1. For month 2 and 3, a brief weekly assessment (Hamilton Rating Scale for Depression-17 score) will be conducted in which it will be determined if they will receive 0, 1 or 2 sessions in the week. For month 4 and 5, a bimonthly assessment (Hamilton Rating Scale for Depression-17 score) will be conducted in which it will be determined if they will receive 0, 1 or 2 sessions over the two weeks. For month 6, one brief assessment (Hamilton Rating Scale for Depression-17 score) will be conducted in which it will be determined if they will receive 0, 1 or 2 sessions in the month.

ELIGIBILITY:
Inclusion Criteria:

1. voluntary and competent to consent to study,
2. female or male aged 18 years old or older,
3. can speak and read English and/or French
4. primary and/or predominant diagnosis of major depressive episode without psychotic features in the current depressive episode (confirmed by a Mini-International Neuropsychiatric Interview),
5. depressive symptoms have not improved after ≥ 1 adequate dose of antidepressant trial in the current depressive episode,
6. moderate symptoms in the current depressive episode as indexed by a score of at least 15 at the 17-item Hamilton Rating Scale for Depression (HRSD-17),
7. have been referred to rTMS treatment by their treating physician, and took a free and informed decision to follow this treatment,
8. are able to adhere to treatment schedule,
9. have received a stable psychiatric medication (including prescribed cannabis) or psychotherapy regimen for at least four weeks prior to entering the trial,
10. have an education-adjusted score of ≥ 24 at the Mini-Mental State Evaluation (MMSE) if are aged ≥ 65.

Exclusion Criteria:

1. current or past (< 3 months) substance (excluding caffeine or nicotine) or alcohol abuse/dependence, as defined in the Diagnostic and Statistical Manual 5th Edition (DSM-5) criteria. Based on the DSM-5 criteria, mild cannabis or alcohol use would be permissible in the past 3 months, moderate to severe would be an exclusion
2. current use of illegal substances or recreational cannabis
3. have a concomitant major unstable medical or neurologic illness (e.g. uncontrolled diabetes or renal dysfunction),
4. organic cause to the depressive symptoms (e.g. thyroid dysfunctions), determined by the referring physician
5. acute suicidality or threat to life from self-neglect,
6. are pregnant or breastfeeding, or thinking of becoming pregnant during course of treatment,
7. have a specific contraindication for TMS (e.g., personal history of epilepsy or seizure, metallic head implant, pacemaker),
8. unwilling to maintain current antidepressant regimen,
9. are taking more than 1 mg of lorazepam or equivalent,
10. any other condition that, in the opinion of the investigators, would adversely affect the participant's ability to complete the study,
11. have failed a course of electroconvulsive therapy (ECT) within the current depressive episode due to the lower likelihood of response to rTMS.If they have had failed ECT in the past, this does not exclude them

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Response - Treatment Phase (Hamilton Rating Scale for Depression-17 score) | Week 6
  Response to treatment will be defined as a > 50% reduction in pre-treatment symptoms severity as measured by the mean Hamilton Rating Scale for Depression-17 score. The minimum value is 0 and the maximum value is 53. A higher score indicates a negative outcome.
Remission - Treatment Phase (Hamilton Rating Scale for Depression-17 Score) | End of treatment phase (week 4 or 6)
  Remission will be defined as a Hamilton Rating Scale for Depression-17 score ≤ 8 The minimum value is 0 and the maximum value is 53. A higher score indicates a negative outcome.
Response - Maintenance Phase (Hamilton Rating Scale for Depression-17 score) | 6 months
  Response to treatment will be defined as a > 50% reduction in pre-treatment symptoms severity as measured by the mean Hamilton Rating Scale for Depression-17 score. The minimum value is 0 and the maximum value is 53. A higher score indicates a negative outcome
Remission - Maintenance Phase (Hamilton Rating Scale for Depression-17 Score) | 6 months
  Remission will be defined as a Hamilton Rating Scale for Depression-17 score ≤ 8 The minimum value is 0 and the maximum value is 53. A higher score indicates a negative outcome.

SECONDARY OUTCOMES:
Response - Treatment Phase (Quick Inventory of Depression Symptomology-Self Report) | Week 6
  Response to treatment will be defined as a > 50% reduction in pre-treatment symptoms severity as measured by the mean the Quick Inventory of Depression Symptomology-Self Report score. The minimum value is 0 and the maximum value is 48. A higher score indicates a negative outcome.
Remission - Treatment Phase (Quick Inventory of Depression Symptomology-Self Report) | End of treatment phase (week 4 or 6)
  Remission will be defined as a Quick Inventory of Depression Symptomology-Self Report score ≤ 6. The minimum value is 0 and the maximum value is 48. A higher score indicates a negative outcome
Response - Maintenance Phase (Quick Inventory of Depression Symptomology-Self Report) | 6 months
  Response to treatment will be defined as a > 50% reduction in pre-treatment symptoms severity as measured by the mean the Quick Inventory of Depression Symptomology-Self Report score. The minimum value is 0 and the maximum value is 48. A higher score indicates a negative outcome.
Remission - Maintenance Phase Quick Inventory of Depression Symptomology-Self Report) | 6 months
  Remission will be defined as a Quick Inventory of Depression Symptomology-Self Report score ≤ 6. The minimum value is 0 and the maximum value is 48. A higher score indicates a negative outcome.

OTHER OUTCOMES:
Cortical Activity - Treatment Phase | Week 6
  TMS-EEG measure of cortical activity (change in pre-treatment TMS-evoked potential amplitude in µV).
Cortical Activity - Maintenance Phase | 6 months
  TMS-EEG measure of cortical activity (change in pre-treatment TMS-evoked potential amplitude in µV).
Resting State Connectivity | 6 months
  Investigate if baseline levels of GABA/Glutamate in the anterior cingulate cortex (ACC) and baseline levels of resting state connectivity between the left dorsolateral prefrontal. cortex (DLPFC) and ACC are linked to therapeutic response, using resting state functional Connectivity between target sites and anterior cingulate cortex (ACC)
Magnetic Resonance Spectroscopy | 6 months
  Baseline levels of gamma-aminobutyric acid (GABA) and Glutamate in the anterior cingulate cortex (ACC)
Cortical Activity in Motor Cortex | 6 months
  Baseline levels excitation and inhibition measured with Transcranial Magnetic Stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tremblay, PhD, Principal Investigator — The Royal Ottawa Mental Health Centre
Locations (1):
- The Royal Ottawa Mental Health Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data collected from this study (IPD) will be de-identified for all parties who have permission to access it. This de-identified data may be shared with other researchers at the Royal's Institute of Mental Health Research. De-identified may be shared with the public only upon request. Please note that all data that has the potential of revealing participants' identity will NOT be used to shared.
Time Frame: De-identified data may become available (upon request) when the study is completed and published (anticipated time frame: the year of 2026)
Access Criteria: De-identified data will be accessible only through the permission of the lead research scientist. All requests must be made and accepted by her.

REFERENCES:
- [Derived] Watson M, Chaves AR, Gebara A, Desforges M, Broomfield A, Landry N, Lemoyne A, Shim S, Drodge J, Cuda J, Kiaee N, Nasr Y, Carleton C, Daskalakis ZJ, Taylor R, Tuominen L, Brender R, Antochi R, McMurray L, Tremblay S. A naturalistic study comparing the efficacy of unilateral and bilateral sequential theta burst stimulation in treating major depression - the U-B-D study protocol. BMC Psychiatry. 2023 Oct 10;23(1):739. doi: 10.1186/s12888-023-05243-4. PMID 37817124